CLINICAL TRIAL: NCT03951129
Title: Determination of Anxiety Levels After Verbal and Video Informing of Hemodialysis Patients Before Hemodialysis Catheter Insertion
Brief Title: Anxiety Levels Before Hemodialysis Catheter Insertion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, huseyin mutlu, Asst. Prof. Dr. Principal Investigator, Aksaray University Training and Research Hospital
Other Study IDs: 587943
Record Dates: First submitted 2019-05-10; First posted 2019-05-15 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Anxiety Levels

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- verbal group: The State-Trait Anxiety Inventory (STAI) and Visual Analogue Scale (VAS) levels after verbal informing before hemodialysis catheter insertion
  Interventions: Procedure: hemodialysis catheter insertion
- verbal and video group: The State-Trait Anxiety Inventory (STAI) and Visual Analogue Scale (VAS) levels after verbal and video informing before hemodialysis catheter insertion
  Interventions: Procedure: hemodialysis catheter insertion

INTERVENTIONS:
Procedure: hemodialysis catheter insertion — The State-Trait Anxiety Inventory (STAI) and Visual Analogue Scale (VAS) scoring will be performed after informing all groups and after the procedure

SUMMARY:
Determination of anxiety levels after verbal and video informing before hemodialysis catheter insertion

DETAILED DESCRIPTION:
Treatment options for end-stage renal patients are renal transplantation, peritoneal dialysis, or hemodialysis, and the majority of these patients live on hemodialysis dependent. The venous access route required for hemodialysis is provided by dialysis catheters until arterio-venous shunts are performed. The aim of this study was to determine the difference between verbal or video-related anxiety levels of patients with hemodialysis and determine which one is better before the hemodialysis procedure is performed.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 -65
* Agree to participate ın the study
* No need for emergency hemodialysis
* No previously known psychiatric disorder
* No history of hemodialysis before
* No history of surgical procedures

Exclusion Criteria:

* Refusing to participate ın the study
* <18 years of age and >65 years
* Need emergency dialysis
* The presence of previously known psychiatric disorder
* Presence of dialysis and catheter
* Presence of a history of surgical procedure
* Lack of information and documents

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study was planned to receive 84 people. The people to be recruited will be divided into groups.
  1. the group will only be informed verbally.
  2. The group will be informed as both verbal and video. State-Trait Anxiety Inventory and VAS score will be made after informing all groups and after Hemodialysis Catheter Insertion
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-06-27 (Estimated); Study Completion 2019-08-27 (Estimated)

PRIMARY OUTCOMES:
The State-Trait Anxiety Inventory (STAI) and Visual Analogue Scale (VAS) levels | 10 minute
  The State-Trait Anxiety Inventory (STAI):To measure via self-report the presence and severity of current symptoms of anxiety and a generalized propensity to be anxious. The STAI has 40 items, 20 items allocated to each of the S-Anxiety and T-Anxiety subscales. Range of scores for each subtest is 20-80, the higher score indicating greater anxiety. A cut point of 39-40 has been suggested to detect clinically significant symptoms for the S-Anxiety scale Visual Analogue Scale (VAS): The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations. Using a ruler, the score is determined by mea-surging the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)

CONTACTS AND LOCATIONS:
Overall Officials: Hüseyin Mutlu, MD, Study Director — Aksaray/Turkey
Locations (1):
- Aksaray Universty, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No